CLINICAL TRIAL: NCT06804135
Title: Systemic and Tumor Immune Response During Pelvic (Chemo)Radiation and/or Brachytherapy for Cervical Cancer (STIRR Cervix Study)
Brief Title: Systemic and Tumor Immune Response During Pelvic (Chemo)Radiation and/or Brachytherapy for Cervical Cancer
Acronym: STIRR
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Professor, Radiation Oncology, Tata Memorial Centre
Other Study IDs: TMH IEC1 No 4591
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cervical Carcinoma
Keywords: Cervical Cancer; Immune System; Radiotherapy; PD-L1 Expression
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Specimen FFPE Tissue Specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cohort A Pelvic RT - Group 1 Radical Cohort: n=20 Fractionation Details = 45Gy/25#
- Cohort A - Group 2 Palliative Arm A: n=20 Fractionation Details = 25Gy/5#
- Cohort A - Group 3 Palliative Arm B: n=20 Fractionation Details = 30Gy/3#
- Cohort B Pelvic + Para aortic RT Group 4: n=20 Fractionation Details = 45Gy/25#
- Cohort C Reirradiation Cohort - Group 5 Proton Therapy: n=10 Fractionation Details = 40Gy/20#
- Cohort C Reirradiation Cohort - Group 6 Photon Therapy: n=10 Fractionation Details = 25-30Gy/5-6#
- Cohort C Reirradiation Cohort - Group 7 SFRT: n=10 Fractionation Details = 45Gy/25#

SUMMARY:
Radiotherapy result in tumor cell death by creating an immune potentiation effect, but can also lead to long lasting immune suppression. Thus the investigators hypothesize that pelvic and/or para-aortic radiotherapy for cervical cancer affects local tumor immunity as well as systemic immune response that may be instrumental for long term cancer cure. The goal of this observational study is to understand the effect of various radiotherapy dose per fraction, total dose and field volumes of radiation on systemic and tumor immune response in cervical cancer. The outcome of the study would be useful in improving the quality of radiation treatment and in reducing disease recurrence and improving survival in patients with cervical cancer.

DETAILED DESCRIPTION:
This study will be performed using blood and tumor material at different time points and available information from blood tests that have been performed prior to initiating chemoradiation in the institution. The proposed sample size is 110 is a convenience based sampling that is based on estimate of people participating in the study during their radiotherapy course. Participants will be allotted in the cohort as per their radiation treatment plan. Collection of blood and tumor tissue material from participants will happen at different time points. These time points will be decided as per the cohort in whom the patient is. The study intends to investigate immunohistochemical (IHC) expression of PD-L1 on baseline and post-treatment tumor biopsy. Furthermore, the study will also investigate expression of immune cells through flow cytometry - fluorescence-activated cell sorter (FACS) at baseline and after RT on blood and tumor tissue sample. The study also intends to capture radiotherapy information - PTV Dose, HRCTV, Mean liver, spleen, Ileocecal junction dose, TRAK values. Using Analysis of Variance (ANOVA) test, all these parameters will be analyzed against their time points in the individual cohorts and also with other cohorts to provide us a better understanding of how pelvic radiotherapy affects our immune system. Furthermore, the investigators will also use Bonferroni correction test to account for multiple statistical comparison. Most of the research studies in cervical cancer that have been published till date do not utilize various aspects of radiotherapy like dose, dose per fraction, field volumes and techniques. This study will represent the first large cohort focusing on all the above mentioned aspects in cervical cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Common Inclusion Criteria:

  1. Age 18 years and above.
  2. Ability to tolerate full course of pelvic radiotherapy+/- chemotherapy +/- brachytherapy.
  3. Ability to understand and willingness to sign an informed consent document.
  4. Should be willing to undergo extra biopsies and blood samples collection for translational research study.

Cohort A:

1. Patients diagnosed with LACC Stage IB2 - IIIC1, as per FIGO 2018 Classification for Radical Cohort.
2. Stage IIIB-IVA where palliative RT is indicated for palliative cohort.
3. No previous irradiation to the pelvis or chemo therapy.

Cohort B:

1. Patients diagnosed with LACC Stage IIIC2, as per FIGO 2018 Classification.
2. No previous irradiation to the pelvis or chemotherapy.

Cohort C:

1. Patients diagnosed with gynecological cancer and presenting with need of infield radiation.
2. Planned for reirradiation.

Exclusion Criteria:

1. Severe medical condition impairing complete treatment delivery.
2. Patients with immunocompromised states or active infection.
3. Patients on immunosuppressive drugs for other medical conditions.
4. Patients who will receive immune checkpoint inhibition (ICI) therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients that are undergoing radiation treatment for primary radiation or reirradiation for cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the systemic immune response in patients undergoing radiotherapy for cervical cancer. | 3 years
  To demonstrate correlation between radiation dose and volume & systemic immune changes during radiotherapy.
To study the multi-time point interaction between radiotherapy for cervical cancer and impact on tumor infiltrating immune cells and PD-L1 expression. | 3 years
  To demonstrate correlation between radiation dose and volume & tumor immune changes during radiotherapy.

SECONDARY OUTCOMES:
To study 3-year disease free survival as a function of baseline and post radiotherapy immune cell composition. | 3 years from last date of treatment and/or to date of reccurrence/relapse
  To determine association of disease-free survival and clinical outcomes with baseline and post radiotherapy immune cell composition.

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No